CLINICAL TRIAL: NCT05905653
Title: Pharmacokinetic Study of STN1012600 Ophthalmic Solution in Healthy Adult Males Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101260007LT
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy Adult Males Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STN1012600 0.002% (Experimental)
  Interventions: Drug: STN1012600 ophthalmic solution 0.002%

INTERVENTIONS:
Drug: STN1012600 ophthalmic solution 0.002% — 1 drop STN1012600 ophthalmic solution 0.002% once daily for 7 days

SUMMARY:
To evaluate the safety and plasma pharmacokinetics of STN1012600 ophthalmic solution 0.002% (1 drop once daily for 7 days) in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who can comply with scheduled visits and the examination and observation as specified in the clinical study protocol

Exclusion Criteria:

* Subjects have a disease and/or abnormal laboratory value which is considered inappropriate from safety evaluation perspective
* Subjects who are inappropriate as participants in this study in the opinion of the investigator or sub investigator

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 1 week, Day 1 and Day 7
  Calculate plasma pharmacokinetic parameters and study pharmacokinetics.

SECONDARY OUTCOMES:
Area Under The Curve From Time Zero to the Last Sampling Time [AUC 0-t] | 1 week, Day 1 and Day 7
  Calculate plasma pharmacokinetic parameters and study pharmacokinetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No